CLINICAL TRIAL: NCT02356354
Title: Study of the Cutaneous Reinnervation After Burn With the Aim of a Better Care of Neuropathic Pain and Pruritus After Healing
Brief Title: Study of the Cutaneous Reinnervation After Burn
Acronym: NERVAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty to recruit all the patients
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RB 14.190 NERVAL
Record Dates: First submitted 2015-01-26; First posted 2015-02-05 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Post-burn Innervation
Keywords: molecular factors; cutaneous innervation; skin biopsy; post-burn scar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin biopsy (Other): On the same patient, a biopsy of post-burn scar is removed. A second one is removed from healthy skin.
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — 2 biopsies are done on the same patient : 20 cutaneous biopsies from post-burn scar and from healthy skin

SUMMARY:
The aim of this study is to understand why the regeneration of the cutaneous sensory nerve fibers is poor in post-burn scar.

The presence or the lack of several molecular factors known to regulate neuronal cell development will be evaluate and compared within biopsies from healthy skin and post-burn scar.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* At least one year back deep burn (2nd and 3rd degrees), and allowing the comparison between the post-burn scar dermatome and the healthy opposite dermatome
* Patients always followed in the service of Plastic surgery of the hospital of Brest
* Informed consent and paper of the patient after information of the objective of the study and the protocol
* Analog Visual scales for pain and/or pruritus (EVA): greater than or equal to 3
* Simple Verbal scales for the pain and/or the pruritus ( EVS): pain / pruritus moderated to intense
* Membership to the Social Security

Exclusion Criteria:

* Allergy to xylocaine
* Non-Caucasian patients
* Treatments having an effect on the pain and/or the pruritus
* Sun or UV exposure several days preceding or following the biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of the differences of expression of genes coding for regulating proteins of the innervation | 6 months
  To evaluate the differences of expression of genes coding for regulating proteins of the innervation on samples of healthy skins and post-burn scar. These biopsies will be removed from post-burn patients (at least one year after burn) and allowing the comparison between conflicting dermatomes: a healthy dermatome and a formerly burned dermatome

SECONDARY OUTCOMES:
Validation of the difference of density of intra-epidermic nerve fibers | 6 months
  To validate the existence of a difference of density of intra-epidermal nerve fibers between the healthy skins and the post-burn scar.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MISERY, Principal Investigator — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France, France